CLINICAL TRIAL: NCT00102141
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study Comparing 3 Continuous Oral Angeliq (Drospirenone 3 mg/17ß-estradiol 1 mg, Drospirenone 2 mg /17ß-estradiol 1 mg, Drospirenone 1 mg /17ß-estradiol 1 mg) Combinations and 17ß-estradiol (1 mg) With Placebo for a Treatment Period of 8 Weeks on Ambulatory and Office Cuff Blood Pressure in Postmenopausal Women With Stage 1 or Stage 2 Essential Hypertension
Brief Title: Effect of Angeliq on Blood Pressure (BP) in Postmenopausal Hypertensive Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 91202; 306743
Record Dates: First submitted 2005-01-21; First posted 2005-01-24 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension; Postmenopause
Keywords: Postmenopausal; vasomotor symptoms; essential hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — estradiol-drospirenone combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891)
- Arm 3 (Experimental)
  Interventions: Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891)
- Arm 4 (Experimental)
  Interventions: Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891)
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2 (Experimental)
  Interventions: Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891)

INTERVENTIONS:
Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891) — Drospirenone 3 mg + 1mg 17ß-estradiol, given as tablets orally once daily in the morning for 8 weeks
  Arms: Arm 1
Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891) — Drospirenone 2 mg + 1mg 17ß-estradiol, given as tablets orally once daily in the morning for 8 weeks
  Arms: Arm 2
Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891) — Drospirenone 1 mg + 1mg 17ß-estradiol, given as tablets orally once daily in the morning for 8 weeks
  Arms: Arm 3
Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891) — 1mg 17ß-estradiol, given as tablets orally once daily in the morning for 8 weeks
  Arms: Arm 4
Drug: Placebo — Placebo, given as tablets orally once daily in the morning for 8 weeks
  Arms: Arm 5

SUMMARY:
The objective of the study is to evaluate the effects of Angeliq on BP over a period of 8 weeks in postmenopausal women who may benefit from hormone replacement therapy (HRT) for the relief of vasomotor symptoms and who have hypertension.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:- Have hypertension- Are currently taking antihypertensive medications- Have had natural menopause at least 1 year prior to screening- Must require hormone therapy in the opinion of the investigator

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2004-04; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Mean change in systolic office blood pressure measured at through | After 8 weeks of treatment
Mean change in 24-hour systolic ambulatory blood pressure measurement (ABPM) | After 8 weeks of treatment

SECONDARY OUTCOMES:
Mean change in diastolic blood pressure measured at through | After 8 weeks of treatment
Mean changes in 24-hour diastolic ABPM | After 8 weeks of treatment
Mean change in daytime systolic ABPM | After 8 weeks of treatment
Mean change in daytime diastolic ABPM | After 8 weeks of treatment
Mean change in nighttime systolic ABPM | After 8 weeks of treatment
Mean change in nighttime diastolic ABPM | After 8 weeks of treatment
Mean change in systolic APBM at through | After 8 weeks of treatment
Mean change in diastolic APBM at through | After 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer